CLINICAL TRIAL: NCT01616719
Title: Evaluation of DTRAX Graft in Patients With Cervical Degenerative Disc Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study was never started due to lack of resources
Sponsor: Providence Medical Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMT002
Record Dates: First submitted 2012-06-07; First posted 2012-06-12 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Cervical Spondylosis; Cervical Radiculopathy; Cervical Degenerative Disc Disease
MeSH Terms: conditions — Spondylosis; Radiculopathy

ARMS (1):
- DTRAX graft (Other)
  Interventions: Device: DTRAX Graft

INTERVENTIONS:
Device: DTRAX Graft — DTRAX Graft is an allograft implant inserted to support spinal fusion.

SUMMARY:
DTRAX Graft is used to relieve nerve pressure in the neck in order to provide relief for Cervical Degenerative Disc Disease. This study is being conducted to determine the effectiveness of the graft, and to find out whether or not it provides better results or faster healing than traditional ways of performing surgery for Cervical Degenerative Disc Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subject diagnosed with DDD in C3-C7, defined as follows:

   * Radiographically (at least one):

     * degenerated disc on MRI;
     * decreased disc height on plain film, CT or MRI; and/or
     * disc herniation, as demonstrated by CT or MRI.
   * Clinically: radicular symptoms (at least one):

     * arm/shoulder pain;
     * decreased reflexes;
     * decreased strength; and/or
     * decreased sensation.
2. Subject has single-level disease, OR multi-level disease demonstrated radiographically, and confirmed to be symptomatic by one of the following methods:

   * Selective nerve root block, OR
   * EMG, OR
   * Distinctive clinical examination.
3. Subject has dynamic stenosis relieved by traction and made worse by a Spurlings maneuver.
4. Subject is 35-80 years of age, inclusive.
5. Subject is unresponsive to 6 weeks conservative, nonoperative treatment, or has the presence of progressive symptoms or signs of nerve root compression in face of combined nonoperative management.
6. Preoperative NDI score of ≥ 30.
7. Preoperative neck pain and arm pain score of ≥ 6 on Neck and Arm Pain Scales.
8. Patient is a male or non-pregnant, non-lactating female.
9. Female patients of child-bearing potential, including those who have had a tubal ligation, but excluding those who have not experienced a menstrual period for at least two years, must have a negative urine pregnancy test at Screening.
10. Patient must voluntarily provide written, informed consent.
11. Subject is able to meet the proposed follow-up schedule.
12. Subject is able to follow the postoperative management program.

Exclusion Criteria:

1. Subject has severe osteopenia, osteoporosis, osteomalacia, spinal metastases, or metabolic bone disease OR the level of BMD is a T score of -2.5 or below OR patient has sustained a vertebral compression or nontraumatic hip or wrist fracture.
2. Subject has overt or active spinal and/or systemic infection.
3. Subject has spondylolisthesis ≥ 3.5mm or rotator subluxation.
4. Subject has cervical myelopathy.
5. Subject has a chronic pain syndrome.
6. Subject has radicular findings with major motor impairment.
7. Subject has a condition that requires postoperative medications that interfere with fusion or the stability of the implant, such as steroids.
8. Subject is mentally incompetent.
9. Subject is a prisoner.
10. Subject is pregnant.
11. Subject abuses alcohol or drugs.
12. Subject has a cervical spinal condition other than symptomatic cervical disc disease requiring surgical treatment at the involved level.
13. Subject has insulin dependent diabetes.
14. Subject has chronic or acute renal failure or prior history of renal disease.
15. Subject has fever at the time of surgery, defined as > 38.5 degrees C.
16. Subject has documented allergy or intolerance to stainless steel, titanium, or a titanium alloy.
17. Subject has received drugs which may interfere with bone metabolism within two weeks prior to the planned date of DTRAX surgery.
18. Subject has history of an endocrine or metabolic disorder known to affect osteogenesis .
19. Subject has had treatment with an investigational therapy within 28 days prior to DTRAX surgery or such treatment is planned during the 16 weeks following implantation of DTRAX Graft.
20. Subject is involved in spinal litigation or Workmen's Compensation claim.
21. Subject is obese, defined as body mass index (BMI) > 35.
22. Patient has psychiatric history, head injury or any other condition, which, in the Investigator's opinion, would prevent the patient from complying with postoperative follow-up visits.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05 (Estimated); Primary Completion 2014-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Gather clinical outcome data on DTRAX Graft. | Baseline throughout 12 months post-operatively
  Clinical outcome data will be collected using the Neck Disability Index (NDI), Visual Analogue Scale (VAS), and a quality of life questionnaire.

SECONDARY OUTCOMES:
Safety information will be evaluated by collecting the type, frequency, severity, device, and procedure-relatedness of adverse events. | Baseline throughout 12 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Bruce McCormack, M.D., Principal Investigator — Neurospine Institute Medical Group; Brian Andrews, M.D., Principal Investigator — Office of Dr. Brian Andrews, Neurosurgery
Locations (2):
- United States (2):
  - Office of Dr. Brian Andrews, Neurosurgery, San Francisco, California
  - Neurospine Institute Medical Group, San Francisco, California